CLINICAL TRIAL: NCT05844293
Title: Single-center, Randomized, Double-blind, Placebo-controlled, Sequential Cohort Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SAD of FXI-GalNAc-siRNA When Administered Subcutaneously to Healthy Subjects.
Brief Title: Single Ascending Dose of FXI-GalNAc-siRNA in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SRN-122-001
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: FXI
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Other): 6 subjects injected with 25 mg dose of FXI-GalNAc-siRNA 2 subjects with Saline
  Interventions: Drug: FXI-GalNAc-siRNA; Other: Placebo
- Cohort 2 (Other): 6 subjects injected with 50 mg dose of FXI-GalNAc-siRNA 2 subjects with Saline
  Interventions: Drug: FXI-GalNAc-siRNA; Other: Placebo
- Cohort 3 (Other): 6 subjects injected with 100 mg dose of FXI-GalNAc-siRNA 2 subjects with Saline
  Interventions: Drug: FXI-GalNAc-siRNA; Other: Placebo
- Cohort 4 (Other): 6 subjects injected with 200 mg dose of FXI-GalNAc-siRNA 2 subjects with Saline
  Interventions: Drug: FXI-GalNAc-siRNA; Other: Placebo
- Cohort 5 (Other): 6 subjects injected with 400 mg dose of FXI-GalNAc-siRNA 2 subjects with Saline
  Interventions: Drug: FXI-GalNAc-siRNA; Other: Placebo

INTERVENTIONS:
Drug: FXI-GalNAc-siRNA — FXI-GalNAc-siRNA solution for injection
  Other Names: FXI-GalNAc-siRNA Solution for Injection
Other: Placebo — Saline

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, PK, and PD of SAD of FXI-GalNAc-siRNA administered SC to healthy subjects.

DETAILED DESCRIPTION:
Phase 1, Single center, randomized, double-blind, sequential cohort study to evaluate safety, tolerability, PK and PD of a single ascending dose of FXI-GalNAc-siRNA when administered subcutaneously in healthy subjects compared with Normal Saline Injection.

The study will include a screening period, treatment period, and a follow-up period.

Five dose cohorts will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all the following criteria will be eligible to participate in the study:

1. Male or female subjects 18 to 55 years of age, inclusive, at the time of signing the informed consent form (ICF).
2. Subjects must be in generally reasonable health with clinically insignificant screening and admission results (medical history, 12-lead electrocardiogram (ECG), physical examination, and laboratory tests), as determined by the Investigator.
3. Subjects must have a body mass index (BMI) ≥ 18 kg/m2 or ≤ 32 kg/m2 at Screening and Day -1 (Admission).
4. Subjects must have aspartate transaminase (AST), alanine transaminase (ALT), total bilirubin (TBIL), alkaline phosphatase (ALP), and glucose within upper limit of normal (ULN) range per reference laboratory reference ranges at Screening and Day -1 (Admission); one repeat laboratory analysis allowed per Investigator discretion.
5. Subjects must have baseline Factor XI plasma levels within normal range as per testing laboratory requirements.
6. Subjects must have prothrombin time (PT) and partial thromboplastin time (PTT) within the ULN range per reference laboratory reference ranges at Screening and Day -1 (Admission); one repeat laboratory analysis allowed per Investigator discretion.
7. Women of childbearing potential must have a negative serum pregnancy test at Screening and negative urine pregnancy test at Day -1 (Admission), must not be actively breastfeeding, or planning to become pregnant during the study, and if not practicing abstinence from heterosexual activity that could result in conception (if this is the preferred and usual lifestyle of the subject), must agree to use 2 approved methods of birth control, during the study and for at least 140 days after study drug administration from the list below:

   1. Condom plus diaphragm with spermicide started at least 28 days prior to dosing.
   2. Condom plus cervical cap or female condom with spermicide started at least 28 days prior to dosing.
   3. Hormonal contraceptives (stable dose for 28 days [4 weeks] prior to Screening) plus condom.
   4. Intrauterine device (in place for 28 days [4 weeks] prior to Screening) plus condom.
   5. Condom plus spermicide.
   6. Partner vasectomy and use of barrier contraception methods (eg, male condom, diaphragm, or sponge with spermicide).
8. Women of nonchildbearing potential must be either surgically sterile (partial/total hysterectomy, bilateral oophorectomy) for at least 6 months confirmed by medical/operative report, or if medical/operative report is not available, confirmed by follicle stimulating hormone [FSH] and 17β-estradiol tests) or > 1 year in the postmenopausal women confirmed by FSH and 17β-estradiol tests.
9. Men must agree to use barrier contraception (condom with a female partner of child-bearing potential who is using oral contraceptives, hormonal patch, implant or injection, intrauterine device or diaphragm with spermicide) and refrain from sperm donation from the day of study drug administration until at least 140 days after study drug administration. Post vasectomy, men must agree to use a barrier method (or partner barrier method) from the day of study drug administration until at least 140 days after study drug administration. Abstinence as a method of contraception is acceptable if it is in line with the preferred and usual lifestyle of the study participant.
10. Subjects must be informed of the nature of the study and must have agreed to and be able to read, review, and sign the study ICF prior to any study-related procedure being performed.

NOTE: If laboratory values are abnormal, tests may be repeated once at Investigator discretion.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Patients with known diagnosis of Hemophilia C, Factor XI deficiency or another known bleeding disorder.
2. Current or previous cancer except superficial forms of non-melanoma skin cancers that have been resolved with clear histology reporting; diabetes or known diagnosis of prediabetes; or any clinically significant cardiovascular (including ECG disturbances or history of rhythm disturbance/abnormality), endocrine, renal, hepatic, gastrointestinal, hematologic, respiratory, dermatological, neurological, psychiatric disorder that could be deemed by the investigator to interfere with study participation, or other disorders that the investigator deems could interfere with study participation.
3. Hypertension, defined as blood pressure > 140/90 mmHg (2 separate readings at least 15 minutes apart if first reading is not within normal range) at Screening and Day -1 (Admission).
4. Hyperlipidemia, defined as:

   1. Cholesterol > 300 mg/dL.
   2. Low-density lipoprotein cholesterol > 190 mg/dL.
   3. And/or triglycerides >500 mg/dL.
5. Hemoglobin A1c (HbA1c) > 6.0% at Screening. Note: Abnormal laboratory values may be repeated once at Investigator discretion
6. Hemoglobin less than 12 g/dL for females and less than 13 g/dL for males or hematocrit outside upper or lower limits of normal range per reference laboratory range at both Screening and Day -1 (Admission).
7. Serum creatinine above ULN per reference laboratory range at both Screening and Day -1 (Admission).
8. Estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73 m2. If GFR value is not supplied by local laboratory, it can be calculated using the Chronic Kidney Disease Epidemiology Collaboration equation at Screening and Day -1 (Admission). One retest of the exclusionary eGFR value is allowed at the discretion of the Investigator.
9. Unwillingness to abstain from alcohol for 72 hours prior to dosing through the EOS Visit (or ET).
10. Use of prescription or nonprescription drugs (excluding hormonal contraceptives), if clinically applicable, including vitamins, supplements, herbal preparations, and medicines that prolong Q wave interval (QT)/ Q wave interval corrected (QTc) within 7 days or 5 times longer than the half-life (whichever is longer) prior to the study drug administration through the EOS Visit (approximately 140 days) or at ET.
11. Blood donation within 56 days or plasma donation within 10 days prior to dosing.
12. Use of live or non-live vaccine (except SARS-CoV-2 and influenza) within 30 days prior to the first dose of study drug or an intention to receive such a vaccine at any time during the study.
13. Received an investigational agent in another clinical study within 30 days prior to the first dose of study drug, or within 10 times longer than the half-life of the compound with which the subject was treated, whichever is longer.
14. Positive results of any of the virology tests (human immunodeficiency virus [HIV test], hepatitis B virus [HBsAg test] or hepatitis C virus [hepatitis C antibody test]).
15. Diagnosed to be SARS-CoV-2 positive based on study center SARS-CoV-2 testing guidelines on Day -1.
16. Personal or family history of vascular aneurysms and disorders.
17. Personal or family history of long QT syndrome.
18. Corrected QT interval using Fridericia's formula (> 450 msec) based on the average of triplicate ECGs.
19. History of active alcoholism or active drug abuse as that would impair the ability of a subject to participate in the study.
20. Positive urine drug or breath alcohol screen at Screening or Day -1 (Admission) and at all visits after confinement, verbal confirmation of compliance.
21. Any condition that, in the opinion of the Investigator, would complicate or compromise the study data or the well-being of the subject.

NOTE: If laboratory values are abnormal, tests may be repeated once at Investigator discretion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Maximum peak concentration | 145 days
  Individual plasma concentration data of FXI-GalNAc-siRNA will be used to determine Maximum peak concentration.
Time to maximum concentration. | 145 days
  Individual plasma concentration data of FXI-GalNAc-siRNA will be used to determine time to maximum concentration.
Apparent terminal elimination rate constant. | 145 days
  Individual plasma concentration data of FXI-GalNAc-siRNA will be used to determine apparent terminal elimination rate constant.
Half life | 145 days
  Individual plasma concentration data of FXI-GalNAc-siRNA will be used to determine half life.
Area under the curve | 145 days
  Individual plasma concentration data of FXI-GalNAc-siRNA will be used to determine area under the plasma concentration-time curve from 0 to the last quantifiable plasma concentration.
Area under the curve from 0-infinity | 145 days
  Individual plasma concentration data of FXI-GalNAc-siRNA will be used to determine area under the curve from time 0 to infinity.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Lebel, MD, Study Director — Chief Medical Officer
Locations (2):
- BioPharma, Creve Coeur, Missouri, United States
- BioPharma, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No